CLINICAL TRIAL: NCT02743988
Title: Influence of Oxygen Target Range on Intermittent Hypoxemia in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Manuel Schmid, MD, University of Ulm
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ULMNEONIRS05
Record Dates: First submitted 2016-04-07; First posted 2016-04-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Intermittent Hypoxemia; Apnea of Prematurity
Keywords: cerebral oxygenation; NIRS; near-infrared spectroscopy; bradycardia; hypoxemia; cerebral perfusion; cardiac output; apnea; desaturation; oxygen saturation target range
MeSH Terms: conditions — Apnea; Bradycardia; Hypoxia | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low target range (Experimental): Low oxygen saturation target range: SpO2 85-89%
  Interventions: Drug: Oxygen
- High target range (Active Comparator): High oxygen saturation target range: SpO2 91-95%
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Adapt inspired oxygen to achieve desired SpO2 target range

SUMMARY:
In this randomized crossover trial, preterm infants with intermittent hypoxemia and need for supplemental oxygen will be randomized to either Sequence of two different oxygen target ranges (low: 85-89%; high: 91-95%) for a total duration of 19 hours. Cerebral oxygenation, cardiac output, arterial oxygenation and heart rate will be measured continuously. Primary outcome is time with arterial oxygen saturation < 80%.

ELIGIBILITY:
Inclusion Criteria:

* preterm infant < 29 weeks gestation
* at least 8 hypoxemic events during 8 hours
* requires supplemental oxygen to achieve high SpO2 target range
* parental consent given

Exclusion Criteria:

* congenital life-threatening malformation
* fatal outcome expected
* airway malformation
* higher grade intraventricular bleeding (grade III or IV according to LA Papile)
* posthaemorrhagic hydrocephalus
* life-threatening disease at the time of study entry

Ages: 21 Days to 42 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Duration SpO2 < 80% | during 16 hours of measurement

SECONDARY OUTCOMES:
Cerebral tissue oxygen saturation as measured by NIRS | during 16 hours of measurement
  Area under threshold
Arterial SpO2 as measured by pulse oxymetry | during 16 hours of measurement
  Area under 80%
Heart rate as measured by ECG | during 16 hours of measurement
  Area under 80/min
cerebral and visceral fractional oxygen extraction as measured by NIRS | during 16 hours of measurement
Cardiac output as measured by Cardiovelocimetry | during 16 hours of measurement
Number of hypoxemic and / or bradycardic events | during 16 hours of measurement
Visceral tissue oxygen saturation as measured by NIRS | during 16 hours of measurement
  Area under threshold

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center, Ulm University, Ulm, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No